CLINICAL TRIAL: NCT00683917
Title: A Multi-center, Active Controlled, Pharmacokinetic, Safety and Efficacy Study of Proellex in Pre-Menopausal Women With Symptomatic Uterine Fibroids to Assess Persistence of Response
Brief Title: Pharmacokinetics, Safety and Efficacy Study of Proellex in Pre-menopausal Women With Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Repros stopped the study for safety and FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZPU-202
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate; Leuprolide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Proellex 25 mg (Experimental): Proellex 25 mg
  Interventions: Drug: Proellex 25 mg
- Proellex 50 mg (Experimental): Proellex 50 mg
  Interventions: Drug: Proellex 50 mg
- Lupron (Active Comparator): Lupron Depot
  Interventions: Drug: Lupron Depot

INTERVENTIONS:
Drug: Proellex 25 mg — Proellex 25 mg, 1 capsule daily for 4 months
  Other Names: Telapristone acetate
  Arms: Proellex 25 mg
Drug: Proellex 50 mg — Proellex 50 mg, 2 capsules daily for 4 months
  Other Names: Telapristone acetate
  Arms: Proellex 50 mg
Drug: Lupron Depot — Lupron 3.75 mg monthly intramuscular injections for 4 months
  Other Names: Leuprolide acetate
  Arms: Lupron

SUMMARY:
PK of 25 mg and 50 mg Proellex® administered once daily (QD) over a 4-month period.

DETAILED DESCRIPTION:
The primary objective is to evaluate the pharmacokinetics (PK) of 25 mg and 50 mg Proellex® administered once daily (QD) over a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects between the ages of 18 and 45 years with body mass index (BMI) between 18 and 35 mg/kg2 inclusive
* Surgical interventions for uterine fibroids (e.g., hysterectomy, myomectomy, or uterine arterial embolization) must not be planned or anticipated during the study
* Subject must have the following uterine fibroid-associated symptom: history of excessive menstrual bleeding
* Regular or steady menstrual cycle lasting from 24 to 36 days
* Willing to comply with all study procedures including the endometrial biopsies and PK blood draws for all visits including follow-up visits
* Subject must agree to use a medically acceptable and effective non-hormonal, double barrier birth control method throughout the study and for 30 days following the end of the study or discontinuation of study drug

Exclusion Criteria:

* Documented endometriosis or active pelvic inflammatory disease
* History of alcohol and/or drug abuse
* Any history or diagnosis of gynecological cancer or cervical dysplasia
* Use of an IUD
* Use of prohibited concomitant medications:

  * Use of Depo-Provera must cease 10 months prior to first dose of study drug
  * Use of GnRH agonists (e.g., Lupron®) must cease 4 months prior to first dose of study drug and Lupton® Depot 8 months prior to the first visit
* Known active infection with HIV; Hepatitis A, B or C; gonorrhea; or chlamydia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAs, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (4):
- United States (3):
  - Physician Care Clinical Research, Sarasota, Florida
  - Advances in Health, Inc., Houston, Texas
  - West Houston Clinical Research Services, Houston, Texas
- Centro de Estudios Cientificos y Clinicos Pharma, S.A. de C.V. (CECYC-Pharma), Mexico City, Federal District, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Proellex All Groups: Proellex 25 mg: Proellex 50 mg, placebo, 1 capsule daily for 4 months Study prematurely terminated, no further data available
Period: Overall Study
Arm/Group | Proellex All Groups
Started | 10
Completed | 0
Not Completed | 10
Not completed — Study prematurely terminated | 10

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Proellex 25 mg | Proellex 50 mg | Lupron | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is the PK Characteristics of 25 mg and 50 mg Proellex.
Time Frame: 4 months
Population: Study prematurely terminated
Arm/Group | Proellex 25 mg | Proellex 50 mg | Lupron
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: No adverse event data is available.
Arm/Group | Proellex 25 mg | Proellex 50 mg | Lupron
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights